CLINICAL TRIAL: NCT06847113
Title: MAXIMAL and SELF-SELECTED WALKING SPEED AFTER KNEE ARTHROPLASTY
Brief Title: Maximal and Self-selected Walkingspeed After Knee Arthroplasty - a Prospective Cohort Study
Acronym: LOVKNEE
Status: Recruiting | Type: Observational
Sponsor: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 764176
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Knee Arthroplasty, Total
MeSH Terms: interventions — Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Persons scheduled for knee arthroplasty: Age 55 or over, scheduled for primary uni or total knee arthroplasty, able to walk indepentdently with or without walkingaids, living in the eastern part of Norway within 1-2 hours commute from Oslo, able understand Norwegian for instructions and filling out forms,
  Interventions: Other: Physical function

INTERVENTIONS:
Other: Physical function — Observe walking speed, both maximal and self-selected, over a 12-months period after knee arthroplasty

SUMMARY:
The purpose of this prospective study is to explore whether maximal and self-selected walking speed in individuals with knee arthroplasty is a useful and applicable clinical measure that can provide new insights into physical function after prosthetic surgery. We will examine the progression of walking speed and other measures of physical function, and investigate if walking speed can predict postoperative function. Individuals over 55 years, scheduled for knee arthroplasty will be invited to participate. Standardized functional tests such as walking speed, sit to stand and one legged stance along with patient reported outcomes will be assessed preoperatively, three months and 12 months after surgery. The study may provide useful knowledge that can be aplied clinically in the assessment and follow-up of this patient group.

ELIGIBILITY:
Inclusion Criteria: age 55 +, living in or near the city of Oslo (up to appox 2 hours commute), sceduled for primary knee arthroplasty, able to walk independently with or without walking aids, understand and speak Norwegian sufficently to take instructions and respond to questionnaires

Exclusion Criteria:

Other reasons than osteoarthritis for knee arthroplasty, revision due to infection or failure, arthroplasty in the same or other limb during the 12 months time period, severe neurological or ohter types of disease that affects walking (e.g MS; parkinsonism, hemiplegiea)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with knee osteoarthritis scheduled for knee arthroplasty at Lovisenberg Diaconal Hospital who meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 3 and 12 months in means in maximal and self-selected walking speed walikgn | Baseline, 3 months and 12 months after surgery
  Walking speed will be measured by 10 meter self-selected and maximal walking speed, respectively. Participant will perform two repetitions of self-selected walking speed, followed by two repetitions of maximal walking speed. Mean, measured by meters per seconds, will be calculated onboth of the two different walking speeds.

SECONDARY OUTCOMES:
Sit-to-stand | Baseline, 3 months and 12 months after surgery
  Lower extremity strength will be measured by 30 sec sit to stand. Number of standing up in 30 seconds will be counted and recorded
One legged stance | Baseline, 3 months and 12 months after surgery
  Balance will be measured by one legged stance. The participant will perform the test by standing on one leg and the other in 90 degrees flexion of the hip and knee, hands on hips. The test will be performed twice, with the non-affected leg to be tested first. The best of the two scores for each leg will be recorded.
Knee specific function and pain | Baseline and 12 months
  Pain and function in the knee will be measured by the patient reported form KOOS which includes 42 questions evaluating pain and function in different activities in daily life the last week.
EQ5D- Health-related quality of life | Baseline and 12 months after surgery
  Measures self-reported health-related quality of life.

OTHER OUTCOMES:
Physical activity | Baseline and 12 months after surgery
  To measure physical activity UCLA activity score will be applied. UCLA is a simple scale from 1 to 10 where the participant mark the level that suits their level of activity best. 1 is the lowest, 10 the highest score.

CONTACTS AND LOCATIONS:
Locations (1):
- Lovisenberg Diaconal Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No